CLINICAL TRIAL: NCT02258724
Title: Swiss National Registry of Grown up Congenital Heart Disease (GUCH) Patients
Brief Title: Swiss National Registry of Grown up Congenital Heart Disease Patients
Acronym: GUCH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 180/13
Record Dates: First submitted 2014-09-24; First posted 2014-10-07 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect
Keywords: Adult; Registry; Grown-up congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to successes in the last decades in pediatric heart surgery and cardiology, 90-95% of the children with congenital heart disease reach adult age.This results in an increasing number of adults or "grown-ups" with congenital heart disease (ACHD or GUCH patients) that require special health care organization and training programmes. Long term complications of these GUCH patients and optimum treatment strategies are still poorly known. The aim of this registry is to collect quantitative and qualitative data regarding GUCH patients treated in specialised centres in Switzerland.

DETAILED DESCRIPTION:
The SWISS GUCH registry will capture epidemiologic data, diagnosis, type of earlier treatment / intervention and cardiac complications. Following each visit, the cardiac complications will be captured as well as the mortality.

Every GUCH patient coming for a visit in one of the specialized organisation participating to the registry will be asked to participate. After signing the informed consent form, the patient data will be coded and captured in a web-based data base (secuTrial®).

Pooling the data from the different centres will enable a nation wide register to be established. More robust data on the size and composition of the GUCH population will be obtained. Also long term prognosis of specific patient group will be derived.

ELIGIBILITY:
Inclusion Criteria:

Adult (above 18 years of age) with congenital heart disease, treated in one of the Swiss centre with specialized organisation for GUCH patients.

Signed informed consent. Patients with trisomy 21: the parents or legal guardian will have to give the consent.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GUCH patient treated in one of the Swiss centre with specialized organisation GUCH (University Hospital Basel, University Hospital Zurich, University Hospital Lausanne, University Hospital Geneva, Canton Hospital StGallen).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-09; Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year and yearly up to 20 years

SECONDARY OUTCOMES:
Cardial complications | 1 year and yearly up to 20 years
  Requiring in-patient hospitalisation, strokes, re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tobler, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (6):
- Switzerland (6):
  - Basel University Hospital, Basel
  - Bern University Hospital Inselspital, Bern
  - Hôpitaux Universitaires de Genève HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

REFERENCES:
- [Background] Moons P, Bovijn L, Budts W, Belmans A, Gewillig M. Temporal trends in survival to adulthood among patients born with congenital heart disease from 1970 to 1992 in Belgium. Circulation. 2010 Nov 30;122(22):2264-72. doi: 10.1161/CIRCULATIONAHA.110.946343. Epub 2010 Nov 22. PMID 21098444
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Derived] Arslani K, Roffler N, Zurek M, Greutmann M, Schwerzmann M, Bouchardy J, Rutz T, Ehl NF, Jost CA, Tobler D; SACHER Investigators. Patterns of Incidence Rates of Cardiac Complications in Patients With Congenital Heart Disease. Can J Cardiol. 2018 Dec;34(12):1624-1630. doi: 10.1016/j.cjca.2018.09.010. Epub 2018 Sep 29. PMID 30527151